CLINICAL TRIAL: NCT06213480
Title: Supplementation With a Next-Generation Synbiotic in Individuals With Overweight or Obesity: A Triple-Blinded Randomized Controlled Clinical Trial
Brief Title: Next-Generation Synbiotic in Individuals With Overweight or Obesity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Texas Christian University (Other)
Collaborators: Pendulum Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2023-345
Record Dates: First submitted 2023-12-20; First posted 2024-01-19 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: Sixty participants will be randomized into one of two groups: 1) 3-day antibiotic plus placebo for 3 months, or 2) 3-day antibiotic plus symbiotic for 3 months.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a triple-blind study. Participants, the research staff, the PI, and the biostatistician will be all blinded. A university staff person who does not belong to the research team or the funding agency but has been CITI certified and approved by the IRB will hold the key of the assignment key.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Synbiotic Group (Experimental): They will receive a 3-day antibiotic (Vancomycin 500 mg/3 times/day), followed by a 3-month symbiotic. The synbiotic that will be used in this trial contains the oligosaccharide-degrading probiotics, Akkermansia muciniphila and Bifidobacterium infantis; butyrate producers such as Clostridium beijerinckii, Anaerobutyricum hallii, and Clostridium butyricum; and chicory-derived inulin, a prebiotic dietary fiber.
  Interventions: Dietary Supplement: Synbiotic Group
- Placebo Group (Placebo Comparator): They will receive a 3-day antibiotic (Vancomycin 500 mg/3 times/day), followed by a 3-month placebo.
  Interventions: Other: Placebo Group

INTERVENTIONS:
Dietary Supplement: Synbiotic Group — WBF-038: Noninfectious and nonhazardous lyophilized commensal bacteria (probiotics). Contains no genetically modified organisms (GMOs) and contains no animal ingredients or by-products, and were originally isolated from human sources. The (probiotic) strains are grown in a FDA registered food facility, adhering to Good Manufacturing Practice (GMP) conditions.
  Probiotic Ingredients:
  Clostridium butyricum WBSTR-0006, Clostridium beijerinckii WB-STR-0005, Anaerobutyricum hallii WB-STR-0008, Akkermansia muciniphila WBSTR-0001, and Bifidobacterium infantis
  The product also contains: Chicory inulin and oligofructose (prebiotic fiber), hypromellose (vegetarian capsule), fruit & vegetable juice (coloring agent), magnesium stearate and silica (flow agent for encapsulation)
  Other Names: The utilized synbiotic is Pendulum Glucose Control
  Arms: Synbiotic Group
Other: Placebo Group — Ingredients: Chicory inulin and oligofructose (prebiotic fiber, hypromellose (vegetarian capsule), fruit & vegetable juice (coloring agent), magnesium stearate and silica (flow agent for encapsulation).
  Other Names: Placebo
  Arms: Placebo Group

SUMMARY:
This study plans to evaluate the effect of consuming a symbiotic (probiotic + prebiotic) for 3 months on body weight, body composition, glucose sensitivity, and psychological parameters, as well as on gut and blood microbial composition. Synbiotic consumption is preceded by a 3-day antibiotic course to help ensure the opening of new niches (houses) for the upcoming beneficial bacteria.

DETAILED DESCRIPTION:
This is a triple-blinded, randomized clinical trial in which participants will be allocated to one of two groups: 1) 3-day antibiotic followed by synbiotic consumption for 3 months or 2) 3-day antibiotic followed by placebo consumption for 3 months.

Blood and stool samples will be collected before the antibiotic, and before and after the symbiotic intervention in both groups.

Gut microbial composition will be analyzed through whole genome sequencing and blood microbial composition through 16S rRNA.

Glucose sensitivity will be measured through fasting glucose, fasting insulin, and HbA1c.

Body composition through DXA and BodPod will be measured before and after the symbiotic intervention.

Psychological questionnaires such as the Beck Anxiety and the Beck Depression Inventories, as well as the RED-9 questionnaire to respectively measure anxiety, depression, and food cravings, will be applied before and after the symbiotic intervention.

ELIGIBILITY:
Inclusion Criteria:

* be between 18-50 years of age
* have a BMI between 25.0-40.0

Exclusion Criteria:

* are following a vegetarian, vegan, carnivore, or keto diet
* currently taking metformin, GLP-1 agonists, insulin, or fiber
* have taken antiacids, laxatives, probiotics, or medication that affects your immune system in the past month
* pregnant, planning pregnancy during the study period, or lactating
* have a history of inflammatory bowel disease, colon cancer, or chronic polyps
* have been diagnosed with type 1 or type 2 diabetes
* have active cancer
* are currently participating in a weight loss intervention (dietetic or medication)
* have used antibiotics, antifungals, or antivirals in the past 3 months
* have had a history of recent (within 30 days) diarrhea illness
* have a known allergy to any component of the study product
* have had an acute inflammatory infection or inflammatory condition in the past 4 weeks
* have had >10% weight variation in the past 6 months
* have had any bariatric surgery

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-01-10 (Estimated); Primary Completion 2024-12-20 (Estimated); Study Completion 2025-05-20 (Estimated)

PRIMARY OUTCOMES:
Total Body Fat Mass through DXA (percentage) | These analyses will take place right before and right after the 3-month synbiotic/placebo intervention.
  We will measure body fat mass by using DXA analysis.
Total Body Fat Mass through BodPod (percentage) | These analyses will take place right before and right after the 3-month synbiotic/placebo intervention.
  We will measure body fat mass by using BodPod analysis.
Fat Mass to Height (kg/m2) | These analyses will take place right before and right after the 3-month synbiotic/placebo intervention.
  We will measure body fat mass by using DXA analysis.
Fat Mass (kg) | These analyses will take place right before and right after the 3-month synbiotic/placebo intervention.
  We will measure body fat mass by using BodPod analysis.
Body Lean Mass to Height (kg/m2) | These analyses will take place right before and right after the 3-month synbiotic/placebo intervention.
  We will measure body lean mass by using DXA analysis.
Fat Free Mass (%) | These analyses will take place right before and right after the 3-month synbiotic/placebo intervention.
  We will measure body lean mass by using BodPod analysis.
Fat Free Mass (Kg) | These analyses will take place right before and right after the 3-month synbiotic/placebo intervention.
  We will measure body lean mass by using BodPod analysis.
Visceral Fat Volume (cm3) | These analyses will take place right before and right after the 3-month synbiotic/placebo intervention.
  We will measure body visceral mass by using DXA and BodPod analysis.
Visceral Fat Mass (grams) | These analyses will take place right before and right after the 3-month synbiotic/placebo intervention.
  We will measure body visceral mass by using DXA and BodPod analysis.
Fasting Glucose (mg/dL) | Blood samples will be taken before the antibiotic, before the synbiotic/placebo, and right after the 3-month synbiotic/placebo intervention.
  We will measure fasting glucose after a 12h fast.
Fasting Insulin (mIU/L) | Blood samples will be taken before the antibiotic, before the synbiotic/placebo, and right after the 3-month synbiotic/placebo intervention.
  We will measure fasting insulin after a 12h fast.
HbA1c (%) | Blood samples will be taken before the antibiotic, before the synbiotic/placebo, and right after the 3-month synbiotic/placebo intervention.
  We will measure HbA1c after a 12h fast.
Anxiety (number in 0-63 scale) | These questionnaires will be applied right before and right after the 3-month synbiotic/placebo intervention.
  We will measure anxiety by using the Beck Anxiety inventory. The higher the number, the higher the anxiety levels.
Depression (number in 0-63 scale) | These questionnaires will be applied right before and right after the 3-month synbiotic/placebo intervention.
  We will measure depression by using the Beck Depression inventory. The higher the number, the higher the depression.
Food cravings (number in 0-52 scale) | These questionnaires will be applied right before and right after the 3-month synbiotic/placebo intervention.
  We will measure food cravings by using the Reward-based Eating Drive questionnaire (RED-9). The higher the number, the higher the cravings.
Gut Microbial Composition (depending on funding availability at the time of analysis) | Stool samples will be collected right before the antibiotic, right before the synbiotic/placebo intervention, and right after the 3-month synbiotic/placebo intervention.
  We plan to measure gut microbial composition by performing whole metagenome sequencing previously stored in Zymo stool collection tubes.
Blood Microbial Composition (depending on funding availability at the time of analysis) | Blood samples will be collected right before the antibiotic, right before the synbiotic/placebo intervention, and right after the 3-month synbiotic/placebo intervention.
  We plan to measure blood microbial composition by performing 16S rRNA in blood samples previously stored in Zymo blood collection tubes.
Body Weight (kg) | Measurements will take place at each of the 3 visits: right before the antibiotic, right before the synbiotic/placebo, and right after the 3-month synbiotic/placebo intervention.
  Body weight will be measured with a calibrated scale.
Body Height (meters) | Measurement will take place at the first visit.
  Body height will be measured with a stadiometer.

CONTACTS AND LOCATIONS:
Overall Officials: Elisa Marroquin, Ph.D., Principal Investigator — Texas Christian University

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant-level data can be shared only after authors and co-authors have published the material of their interest.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available only after authors and co-authors have published the material of their interest.
Access Criteria: Not available at this point. Recruitment has not started.

REFERENCES:
- [Background] Depommier C, Everard A, Druart C, Plovier H, Van Hul M, Vieira-Silva S, Falony G, Raes J, Maiter D, Delzenne NM, de Barsy M, Loumaye A, Hermans MP, Thissen JP, de Vos WM, Cani PD. Supplementation with Akkermansia muciniphila in overweight and obese human volunteers: a proof-of-concept exploratory study. Nat Med. 2019 Jul;25(7):1096-1103. doi: 10.1038/s41591-019-0495-2. Epub 2019 Jul 1. PMID 31263284
- [Background] Perraudeau F, McMurdie P, Bullard J, Cheng A, Cutcliffe C, Deo A, Eid J, Gines J, Iyer M, Justice N, Loo WT, Nemchek M, Schicklberger M, Souza M, Stoneburner B, Tyagi S, Kolterman O. Improvements to postprandial glucose control in subjects with type 2 diabetes: a multicenter, double blind, randomized placebo-controlled trial of a novel probiotic formulation. BMJ Open Diabetes Res Care. 2020 Jul;8(1):e001319. doi: 10.1136/bmjdrc-2020-001319. PMID 32675291

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-12-18): https://cdn.clinicaltrials.gov/large-docs/80/NCT06213480/Prot_SAP_000.pdf
  • Informed Consent Form (2023-12-19): https://cdn.clinicaltrials.gov/large-docs/80/NCT06213480/ICF_001.pdf